CLINICAL TRIAL: NCT04607213
Title: Comparison of Rotation- Advancement and Straight-line Methods for Repairing of Unilateral Cleft Lip (Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Rotation-advancement and Straight-line Surgical Approaches in Repairing Unilateral Cleft Lip Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cleft lip_00010556
Record Dates: First submitted 2020-10-16; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Unilateral Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advancement-rotation approach (Active Comparator)
  Interventions: Procedure: Advancement-rotation approach based on Millard' for repairing lip defect.
- Straight-line approach (Experimental)
  Interventions: Procedure: Straight-line approach

INTERVENTIONS:
Procedure: Advancement-rotation approach based on Millard' for repairing lip defect. — patients were treated using Millard technique is the downward rotation of the medial part of the flap, and lateral advancement of the flap to close and fill the defect. if more lip height is needed; "cut- as- you-go" by adding a back-cut incision at the end of his rotation incision down toward the philtral ridge of non-clefted side. Moreover; C-flap is used to close nasal sill.
  Arms: Advancement-rotation approach
Procedure: Straight-line approach — patients were treated using Straight-Line design based on Fisher modification. C-shaped flap extend from the proposed nasal sill to the origin of philtral column of medial flap as a straight incision to the planned top of the cupid's bow. In addition, to the previous mentioned incision, small inlate incision is needed to length the cleft side on the medial flap.
  On the other hand, on the lateral flap; two connected triangular incisions are used; one on the vermillion border at Noordhoff's point. And the other one just above the cutaneous margin to improve aesthetic outcome and diminish formed scar.
  Arms: Straight-line approach

SUMMARY:
compare different effects of Rotation-advancement based on the Millard technique and Straight-line based on Fisher modification as surgical approaches in repairing lip defect of unilateral cleft lip patients.

DETAILED DESCRIPTION:
Twelve participants with unilateral cleft lip equally divided into two groups. Both groups were photographed preoperative and postoperative. The Control group treated using (Rotation-advancement) based on the Millard technique; and the test group treated using (Straight-line) technique based on Fisher modification.

ELIGIBILITY:
Inclusion Criteria:

* Have complete unilateral cleft lip
* from birth to 4 years old

Exclusion Criteria:

* syndromic cleft patient

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
change in vertical and horizontal lip length | at 3rd, 6th months
  Measuring vertical and horizontal lip length of the constructed philtral ridge by caliper
change in lip defect | at 1st, 3rd and 6th months
  repaired lip is evaluated by direct visual inspection for the patient evaluation.

SECONDARY OUTCOMES:
change in degree of labial scaring | at 3rd, 6th months
  Using a five-point scale based on Asher-McDade scoring system:
  (very good, good, fair, poor, very poor on a scale of 1-5, where 5 represents very poor and 1 represent very good).
change in nasal symmetry | at 3rd, 6th months
  measuring total nasal width and nostril width by caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt